CLINICAL TRIAL: NCT00090896
Title: A Phase I, Open Label, Study To Evaluate The Safety And Immune Function Effects Of CP-675,206 In Combination With MART-1 Peptide-Pulsed Dendritic Cells In Patients With Advanced Melanoma
Brief Title: CP-675,206 (CTLA4-Blocking Monoclonal Antibody) Combined With Dendritic Cell Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed With Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000380840; UCLA-0312023; PFIZER-NRA3670003
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CTLA4-Blocking Monoclonal Antibody (Experimental)
  Interventions: Biological: maximum tolerated dose of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody

INTERVENTIONS:
Biological: maximum tolerated dose of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody

SUMMARY:
RATIONALE: Biological therapies, such as CP-675,206, work in different ways to stimulate the immune system and stop tumor cells from growing. Vaccines may make the body build an immune response to kill tumor cells. Combining CP-675,206 with vaccine therapy may cause a stronger immune response and kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of CP-675,206 when given with vaccine therapy in treating patients with stage III or stage IV melanoma that cannot be removed with surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and maximum tolerated dose of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (CTLA4-blocking monoclonal antibody; CP-675,206) administered with autologous dendritic cells pulsed with MART-1 antigen in patients with unresectable stage III or stage IV melanoma.
* Determine the biological activity and immune effects of this regimen in these patients.

Secondary

* Correlate CTLA4 genotype with safety of this regimen and/or immune response in these patients.
* Determine, preliminarily, the efficacy of this regimen, in terms of clinical benefit rate, in these patients.

OUTLINE: This is an open-label, dose-escalation study of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (CTLA4-blocking monoclonal antibody; CP-675,206).

Patients receive CP-675,206 IV on days 0, 28, 60, and 90 and autologous dendritic cells pulsed with MART-1 antigen intradermally on days 0, 14, and 28. After day 120, patients with stable or responding disease may receive additional doses of CP-675,206 monthly in the absence of disease progression or unacceptable toxicity

Cohorts of 3-6 patients receive escalating doses of CP-675,206 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 3-21 patients will be accrued for this study within 3-10 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cutaneous or mucosal melanoma, meeting criteria for 1 of the following:
* Unresectable stage III disease (locally relapsed unresectable, in-transit lesions, or unresectable draining nodes)
* Stage IV disease, metastatic to 1 of the following sites:

  * Skin, subcutaneous tissues, or distant lymph nodes
  * Lung
  * Other visceral sites with lactic dehydrogenase ≤ 2 times upper limit of normal (unless due to liver stasis)
* De novo metastatic disease allowed provided patient refused any standard or approved stage-appropriate therapy for melanoma
* Measurable disease
* HLA-A2.1 positive (HLA-A*0201 by molecular subtyping)
* MART-1-expressing tumor by reverse transcription polymerase chain reaction or immunohistochemistry
* No symptomatic brain metastases and/or progression of CNS metastases within the past 4 weeks
* Age 18 and over
* Performance status ECOG 0-1 OR
* Karnofsky 70-100%
* HIV negative
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* More than 30 days since prior immunotherapy for metastatic, relapsed, or primary melanoma
* More than 30 days since prior chemotherapy for metastatic, relapsed, or primary melanoma
* More than 4 weeks since prior corticosteroids
* More than 30 days since prior radiotherapy for metastatic, relapsed, or primary melanoma
* More than 30 days since prior surgery for metastatic, relapsed, or primary melanoma.
* More than 30 days since other prior therapy for metastatic, relapsed, or primary melanoma
* More than 14 days since prior anti-infective therapy
* More than 4 weeks since prior immune suppressive therapy (e.g., cyclosporine)

Exclusion Criteria:

* chronic hepatitis B or C
* asthma
* inflammatory bowel disease
* celiac disease
* history of chronic colitis or other chronic gastrointestinal conditions associated with diarrhea or bleeding
* active chronic inflammatory or autoimmune disease, including any of the following:
* Psoriasis
* Rheumatoid arthritis
* Multiple sclerosis
* Hashimoto's thyroiditis
* Addison's disease
* Graves' disease
* Systemic lupus erythematosus
* active infection OR fever over 100° F within the past 3 days
* allergy to study drugs
* pregnant
* symptomatic seizures
* other medical problem that would preclude study participation
* prior melanoma immunotherapy containing MART-1 antigen
* prior anti-T-cell therapy
* prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (CP-675,206)
* organ allografts requiring long-term immune suppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-04; Primary Completion 2008-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Comin-Anduix B, Sazegar H, Chodon T, Matsunaga D, Jalil J, von Euw E, Escuin-Ordinas H, Balderas R, Chmielowski B, Gomez-Navarro J, Koya RC, Ribas A. Modulation of cell signaling networks after CTLA4 blockade in patients with metastatic melanoma. PLoS One. 2010 Sep 15;5(9):e12711. doi: 10.1371/journal.pone.0012711. PMID 20856802